TITLE OF STUDY

Downstream molecular signals of P2Y12 receptors in hyporeactive patients

under clopidogrel treatment

NCT03190005

Unique Protocol ID: TCHIRB-10603117-E

PRINCIPAL INVESTIGATOR

[Name] Chen Yueh Chung

[Department] Taipei City hospital Division of Cardiovascular section

[Address] Ren-Ai Rd, No 10, sec 4, Taipei, Taiwan, ROC

[Phone] 0933060177

[Email] chenyuehchung.tw@yahoo.com.tw

Date: 2018/2/22

**Statistical analysis** 

All numerical variables were depicted in bar charts with mean. Differences

in means between any two groups (hyper- vs. hypo-, normal- vs. hyper-, or

normal vs. hypo-reactive group) were analyzed by Student's t-test. The

Bonferroni test was used to calculate differences between regimens, and reactive

levels. Two-tail and p < 0.05 was considered statistically significant for the

Student's t-test, and two-tail and total p < 0.05 was considered statistically

significant for the Bonferroni test. All plots and statistical analyses were

performed using SAS 9.4 (SAS Institute Inc., Cary, NC, USA) and IBM SPSS 22.